CLINICAL TRIAL: NCT04381845
Title: Immunity and COVID Infections in the Psychiatric Population
Brief Title: Immunity and Infections in the Psychiatric Population
Acronym: COVIDIMMUNOPSY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP200553
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-02

CONDITIONS: COVID; Psychiatric Disorders
Keywords: COVID infection; psychiatric population
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- psychiatric patient (Other): patients who are hospitalized in psychiatric department
  Interventions: Diagnostic Test: COVID19 immunization testing

INTERVENTIONS:
Diagnostic Test: COVID19 immunization testing — serological COVID19 test with confirmation at J15 during hospitalization

SUMMARY:
The main objective of this multicenter cohort study is to determine the degree of COVID19 infection immunization of a population of psychiatric patients.

The secondary objective of this cohort follow-up is to:

1. Clinically characterize COVID patients who are positive for serological testing
2. Assess the socio-demographic, clinical and psychotropic determinants of a COVID diagnosis
3. Immunologically characterize COVID patients who are positive for serological testing
4. Exploring the links between susceptibility to COVID19 and erythrocytic blood groups

DETAILED DESCRIPTION:
All patients accepting to participate will be included in participating psychiatry services and will have a COVID Serological Test for Inclusion with confirmation at J15 including immune-genetics data.

A Comparison of COVID patients versus no COVID patients will be based on a clinical examination (psychiatric, somatic) and blood samples collected at J0 and J15.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Hospitalized in one of the participating psychiatric wards during the inclusion period
* Signed informed consent

Exclusion Criteria:

* Inability to obtain the consent of the patient or legal representative, if applicable
* Patient under safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-10 (Actual); Primary Completion 2023-12-10 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
Number of COVID-positive patients | day 15
  Number of COVID-positive patients, defined by a positive serological test result by immuno-chromatography at inclusion or at 15 days.

CONTACTS AND LOCATIONS:
Overall Officials: Marion LEBOYER, PHD, Principal Investigator — Assistance Publique des Hopitaux de Paris
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No